CLINICAL TRIAL: NCT01103245
Title: Aldosterone and the Metabolic Syndrome: Renin Inhibition Versus Mineralocorticoid Receptor (MR) Antagonism
Brief Title: Aldosterone and the Metabolic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Matt Luther, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 091072; 09CRP2261428 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Diseases; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders
Keywords: Glucose; Insulin
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Insulin Resistance | interventions — Hydrochlorothiazide; aliskiren; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- HCTZ plus ALI 150 then ALI 300 (Active Comparator): Hydrochlorothiazide (HCTZ) 12.5mg daily for 1 month
  then HCTZ 12.5mg daily plus Aliskiren 150 mg (ALI 150) daily for 1 month
  then HCTZ 12.5mg daily plus Aliskiren 300mg ((ALI 300) for 1 month
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Aliskiren 150 mg (ALI 150); Drug: Aliskiren 300 mg (ALI 300)
- HCTZ plus ALI 150 then ALI 150 and SPL 25 (Active Comparator): HCTZ 12.5mg daily for 1 month
  then HCTZ 12.5mg daily plus Aliskiren 150 mg daily for 1 month
  then HCTZ 12.5mg daily plus Aliskiren 150 mg daily and Spironolactone 25mg (SPL 25) daily for one month
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Aliskiren 150 mg (ALI 150); Drug: Spironolactone (SPL 25)
- HCTZ plus SPL 25 then SPL 50 (Active Comparator): HCTZ 12.5mg daily for 1 month
  then HCTZ 12.5mg daily plus Spironolactone 25 mg (SPL 25) daily for 1 month
  then HCTZ 12.5mg daily plus Spironolactone 50 mg daily for one month
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Spironolactone (SPL 25); Drug: Spironolactone 50 mg (SPL 50)
- HCTZ plus SPL 25 then ALI 150 and SPL 25 (Active Comparator): HCTZ 12.5mg daily for 1 month
  then HCTZ 12.5mg daily plus Spironolactone 25 mg daily for 1 month
  then HCTZ 12.5mg daily plus Aliskiren 150 mg daily and Spironolactone 25 mg daily for one month
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Aliskiren 150 mg (ALI 150); Drug: Spironolactone (SPL 25)

INTERVENTIONS:
Drug: Hydrochlorothiazide (HCTZ) — HCTZ 12.5mg daily
  Other Names: HCTZ
Drug: Aliskiren 150 mg (ALI 150) — Aliskiren 150mg daily
  Other Names: Tekturna
  Arms: HCTZ plus ALI 150 then ALI 150 and SPL 25; HCTZ plus ALI 150 then ALI 300; HCTZ plus SPL 25 then ALI 150 and SPL 25
Drug: Spironolactone (SPL 25) — spironolactone 25mg daily
  Other Names: Aldactone
  Arms: HCTZ plus ALI 150 then ALI 150 and SPL 25; HCTZ plus SPL 25 then ALI 150 and SPL 25; HCTZ plus SPL 25 then SPL 50
Drug: Aliskiren 300 mg (ALI 300) — Aliskiren 300mg daily
  Other Names: Tekturna
  Arms: HCTZ plus ALI 150 then ALI 300
Drug: Spironolactone 50 mg (SPL 50) — Spironolactone 50 mg daily
  Other Names: Aldactone
  Arms: HCTZ plus SPL 25 then SPL 50

SUMMARY:
The purpose of this study is to determine the effects of mineralocorticoid receptor (MR) antagonism and renin inhibition on glucose metabolism in humans.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of mineralocorticoid receptor (MR) antagonism and renin inhibition on fasting blood glucose and glucose-stimulated insulin secretion in humans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following conditions will be included in the study:

  1. Ambulatory subjects, 18 to 70 years of age, inclusive
  2. For female subjects, the following conditions must be met:

     1. postmenopausal status for at least 1 year, or
     2. status-post surgical sterilization, or
     3. if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day.
  3. A seated or supine systolic blood pressure greater than 130/85 on three separate measurements at least 15 minutes apart
  4. Metabolic Syndrome as defined by the presence of > 3 of the following:

     1. Hypertension as characterized by having Systolic Blood Pressure > 140 mm Hg and Diastolic Blood Pressure > 90 mm Hg.
     2. Impaired Glucose Tolerance (Fasting Plasma Glucose > 100 mg/dL)
     3. Increased triglyceride level > 150mg/dL
     4. Decreased levels of High-Density Lipoprotein (HDL) cholesterol

        1. For males, less than 30 mg/dL
        2. For females, less than 40 mg/dL
     5. Waist circumference

        1. For males, greater than 40 inches.
        2. For females, greater than 35 inches.

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:

  1. Diabetes type 1 or type 2, a fasting glucose of greater than 110 mg/dL or the use of anti-diabetic medication
  2. Use of hormone replacement therapy
  3. Statin therapy
  4. Pregnancy
  5. Breast-feeding
  6. Cardiovascular disease such as prior myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure [Left Ventricular (LV) hypertrophy acceptable], deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
  7. Treatment with anticoagulants
  8. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack
  9. History or presence of immunological or hematological disorders
  10. Diagnosis of asthma requiring use of inhaled beta agonist >1 time per week
  11. Clinically significant gastrointestinal impairment that could interfere with drug absorption
  12. Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) >1.5 x upper limit of normal range]
  13. Impaired renal function [estimated glomerular filtration rate (eGFR) of <60ml/min] as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dl and age in years:

      eGFR (ml/min/1.73m2)=175 • Scr-1.154 • age-0.203 • (1.212 if black) • (0.742 if female)
  14. Hematocrit <35%
  15. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal antiinflammatory drugs
  16. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
  17. Treatment with lithium salts
  18. History of alcohol or drug abuse
  19. Treatment with any investigational drug in the 1 month preceding the study
  20. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
  21. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
  22. Screening plasma potassium <3.2 mmol/L or use of chronic potassium supplements for the treatment of hypokalemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Luther, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez CE, Shuey MM, Milne GL, Gilbert K, Hui N, Yu C, Luther JM, Brown NJ. Arg287Gln variant of EPHX2 and epoxyeicosatrienoic acids are associated with insulin sensitivity in humans. Prostaglandins Other Lipid Mediat. 2014 Oct;113-115:38-44. doi: 10.1016/j.prostaglandins.2014.08.001. Epub 2014 Aug 28. PMID 25173047

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 of the consented participants did not meet inclusion criteria and did not participate in the study
Groups:
- HCTZ Plus ALI 150 Then ALI 300: Baseline: HCTZ 12.5mg daily for 1 month (Baseline, HCTZ only), then Period 1: HCTZ 12.5mg daily plus Aliskiren 150 mg daily for 1 month (HCTZ + ALI 150), then Period 2: HCTZ 12.5mg daily plus Aliskiren 300mg for 1 month (HCTZ + ALI 300)
- HCTZ Plus ALI 150 Then ALI 150 and SPL 25: Baseline: HCTZ 12.5mg HCTZ daily for 1 month (Baseline, HCTZ only), then Period 1: HCTZ 12.5mg daily plus Aliskiren 150 mg daily for 1 month (HCTZ + ALI 150), then Period 2: HCTZ 12.5mg daily plus Aliskiren 150 mg daily and Spironolactone 25 mg daily for one month (HCTZ + ALI 150 and SPL 25)
- HCTZ Plus SPL 25 Then SPL 50: Baseline: HCTZ 12.5mg HCTZ daily for 1 month (Baseline, HCTZ only), then Period 1: HCTZ 12.5mg daily plus Spironolactone 25 mg daily for 1 month (HCTZ + SPL 25), then Period 2: HCTZ 12.5mg daily plus Spironolactone 50 mg daily for one month (HCTZ + SPL 50)
- HCTZ Plus SPL 25 Then ALI 150 and SPL 25: Baseline: HCTZ 12.5mg HCTZ daily for 1 month (Baseline, HCTZ only) Period 1: HCTZ 12.5mg daily plus Spironolactone 25 mg daily for 1 month (HCTZ + SPL 25) Period 2: HCTZ 12.5mg daily plus Aliskiren 150 mg daily and Spironolactone 25 mg daily for one month (HCTZ + ALI 150 and SPL 25)
Period: Overall Study
Arm/Group | HCTZ Plus ALI 150 Then ALI 300 | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 | HCTZ Plus SPL 25 Then SPL 50 | HCTZ Plus SPL 25 Then ALI 150 and SPL 25
Started | 13 | 7 | 12 | 6
Completed | 10 | 5 | 8 | 6
Not Completed | 3 | 2 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0
Not completed — Inadequate IV access | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: subjects who received drug but dropped out before study outcome measures could be obtained were excluded from final analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | HCTZ Plus ALI 150 Then ALI 300 | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 | HCTZ Plus SPL 25 Then SPL 50 | HCTZ Plus SPL 25 Then ALI 150 and SPL 25 | Total
Number analyzed (Participants) | 13 | 7 | 12 | 6 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 12 | 6 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.8) | 46.8 (8.4) | 44.0 (11.6) | 42.8 (13.8) | 45.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 6 | 1 | 19
  Male | 4 | 4 | 6 | 5 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 7 | 12 | 6 | 38

OUTCOME MEASURES:

1. Primary Outcome: Plasma Insulin
Description: A Hyperglycemic clamp was performed once during each study period to assess glucose stimulated insulin secretion. Glucose is infused intravenously to maintain blood glucose near 200 mg/dL to stimulate insulin secretion. During this time plasma insulin levels were measured and the insulin response is reported as the incremental increase over the first 10 minutes of glucose administration.
Time Frame: at the end of each 1 month study period ( 3 times in total)
Population: 2 participants were excluded from the final analysis because they did not complete any of the Hyperglycemic clamps:1 from the HCTZ plus ALI150 then ALI 300 group and 1 participant from the HCTZ plus SPL 25 then ALI 150 and SPL 25 group.
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | HCTZ Plus ALI 150 Then ALI 300 | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 | HCTZ Plus SPL 25 Then SPL 50 | HCTZ Plus SPL 25 Then ALI 150 and SPL 25
Number analyzed (Participants) | 12 | 7 | 11 | 6
uU/ml
  Baseline, HCTZ Only | 75.4 (82.7) | 50.1 (40.1) | 43.5 (23.9) | 114.0 (93.1)
  HCTZ + ALI 150: number analyzed (Participants) | 12 | 6 | 0 | 0
  HCTZ + ALI 150 | 54.8 (50.2) | 43.3 (33.0) |  |
  HCTZ + ALI 300: number analyzed (Participants) | 10 | 0 | 0 | 0
  HCTZ + ALI 300 | 75.7 (76.6) |  |  |
  HCTZ + ALI 150 and SPL 25: number analyzed (Participants) | 0 | 5 | 0 | 6
  HCTZ + ALI 150 and SPL 25 |  | 69.1 (37.3) |  | 99.9 (32.0)
  HCTZ + SPL 25: number analyzed (Participants) | 0 | 0 | 10 | 6
  HCTZ + SPL 25 |  |  | 53.4 (36.6) | 113.2 (99.7)
  HCTZ + SPL 50: number analyzed (Participants) | 0 | 0 | 8 | 0
  HCTZ + SPL 50 |  |  | 44.3 (18.3) |

2. Primary Outcome: Plasma Glucose
Description: Fasting plasma glucose, measured during hyperglycemic clamp
Time Frame: at the end of each 1 month study period ( 3 times in total)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | HCTZ Plus ALI 150 Then ALI 300 | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 | HCTZ Plus SPL 25 Then SPL 50 | HCTZ Plus SPL 25 Then ALI 150 and SPL 25
Number analyzed (Participants) | 12 | 7 | 11 | 6
mg/dl
  Baseline, HCTZ Only | 108.6 (24.1) | 106.1 (18.1) | 96.4 (10.1) | 102.2 (18.4)
  HCTZ + ALI 150: number analyzed (Participants) | 12 | 6 | 0 | 0
  HCTZ + ALI 150 | 119.7 (39.7) | 105.7 (20.4) |  |
  HCTZ + ALI 300: number analyzed (Participants) | 10 | 0 | 0 | 0
  HCTZ + ALI 300 | 111.4 (25.3) |  |  |
  HCTZ + ALI 150 and SPL 25: number analyzed (Participants) | 0 | 5 | 0 | 6
  HCTZ + ALI 150 and SPL 25 |  | 102.1 (10.9) |  | 107.2 (17.3)
  HCTZ + SPL 25: number analyzed (Participants) | 0 | 0 | 10 | 6
  HCTZ + SPL 25 |  |  | 104.8 (10.7) | 101.7 (11.5)
  HCTZ + SPL 50: number analyzed (Participants) | 0 | 0 | 8 | 0
  HCTZ + SPL 50 |  |  | 105.9 (10.7) |

ADVERSE EVENTS:
Arm/Group | HCTZ Plus ALI 150 Then ALI 300 | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 | HCTZ Plus SPL 25 Then SPL 50 | HCTZ Plus SPL 25 Then ALI 150 and SPL 25
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 6/13 | 7/7 | 5/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCTZ Plus ALI 150 Then ALI 300 (N=13) | HCTZ Plus ALI 150 Then ALI 150 and SPL 25 (N=7) | HCTZ Plus SPL 25 Then SPL 50 (N=12) | HCTZ Plus SPL 25 Then ALI 150 and SPL 25 (N=6)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) — Headache, transient
IV irritation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) — Irritation at IV site
Cramp (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) — muscle cramping
Dizziness or Lightheadedness (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dizziness or lightheadedness, without fall or syncope
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Generalized fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No